CLINICAL TRIAL: NCT05199064
Title: Efficacy of Ultrasound Guided Greater Occipital Nerve Pulsed Radiofrequency Therapy in Chronic Refractory Migraine
Brief Title: Efficacy of Greater Occipital Nerve Radiofrequency for Refractory Migraine Treatment
Status: Completed | Type: Observational
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, derya guner, MD, Tepecik Training and Research Hospital
Other Study IDs: Tepecik TRH
Record Dates: First submitted 2022-01-05; First posted 2022-01-20 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Migraine; Headache Disorders, Primary
Keywords: migraine; ultrasound, greater occipital nerve(GON), radiofrequency
MeSH Terms: conditions — Migraine Disorders; Headache Disorders, Primary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic refractory migraine patients: 25 patients who were diagnosed as having chronic refractory migraine and were refractory to conventional treatments, such as oral medications, GONB,and botulinum toxin injection were evaluated.All patients received pulsed RFtherapy to the GON from the proximal (C2) level in the pain clinic between September 2020 and September 2021.
  Interventions: Other: Ultrasound guided greater occipital nerve (GON) radiofrequency

INTERVENTIONS:
Other: Ultrasound guided greater occipital nerve (GON) radiofrequency — After identifying the GON with ultrasound guidance, a catheter needle (22-gauge 5 cm 5 mm active tip hybrid electrode) is inserted with an in-plane technique from lateral to medial.After visualizing the electrode tip placed close to the right or left GON, a sensory stimulation test is performed using an RF generator (URF-3AP Diros Tecnology Inc.). After the patient reports dysesthesia and a tingling sensation at the occipital area with less than 0.2 V, the PRF treatment is administered at 5 Hz and 5 milliseconds pulsed width for 360 seconds at 45 V under the constraint that the temperature of the electrode tips does not exceed 42°C
  Other Names: GON RF

SUMMARY:
Objective: Ultrasound-guided pulsed radiofrequency therapy can be used on the greateroccipital nerve (GON) in patients with chronic migraine (CM) who are unresponsive to conservative treatments. In this study, we aimed to demonstrate the change in pain intensity, duration of migraine episodes, frequency of attacks,migraine disability, depression,and sleep disturbance scores before and after treatment in patients with CM who underwent ultrasound-guided GON pulsed radiofrequency and the effectiveness of treatment. Patients and methods:The study included 25 patients who were diagnosed as having CMaccording to the International Classification of Headache Disorders III beta version diagnostic criteria. The Migraine Disability Assessment Scale (MIDAS), Beck Depression Inventory(BDI), Pittsburgh Sleep Quality Index (PSQI),and a visual analog scale (VAS) were used on patients before GON pulsed radiofrequency treatment and at post treatment months 1 and 3. Results:The median duration and number of migraine episodes in the post-interventional 1st month and 3rd month were significantly shorter and fewer compared with the pre intervention period (p<0.001). In the comparison with the pre intervention values, all of the scoring concepts, namely the MIDAS, VAS, BDI, and PSQI, revealed a significant drop in the post intervention 1st and 3rd month (p<0.001). Conclusion: In this study, we observed that ultrasound-guided GON pulsed radiofrequency therapy applied at the proximal (C2) level was a safe and effective treatment option.With GON pulsed radiofrequency, we observed a decrease in pain intensity, pain frequency, andduration of episodes, and an improvement in depression symptoms, migraine disability, and sleep disorder scores accompanying chronic migraine.

DETAILED DESCRIPTION:
Design and Study Population:

The ethical approval of the current study was obtained from the Local Ethics Committee of Tepecik Education and Research Hospital. In this study, 25 patients who were diagnosed as having chronic refractory migraine and were refractory to conventional treatments, such as oral medications, GONB,and botulinum toxin injection were evaluated.All patients received pulsed RFtherapy to the GON from the proximal (C2) level in the pain clinic between September 2020 and September 2021. In the current study, patients who were highly likely to have a chronic systemic disease that might be the cause of headache, such as hypertension, were excluded from the study. Additionally, patients who already had other primary headache conditions were also excluded.

To assess the outcomes of the intervention, the patients were evaluated in terms of Beck'sDepression Inventory (BDI) scores,Migraine Disability Assessment Score (MIDAS), visual analog scale (VAS) scores, and Pittsburgh Sleep Quality Index (PSQI) scores.VASsare measurement instruments that try to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. They are often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms such as pain. MIDAS is a brief, self-administered questionnaire designed to quantify headache-related disability over 3 months. The MIDAS score has been shown to have moderately high test-retest reliability in patients with headaches. Psychological symptoms often coexist in patients with migraine. Symptoms of depression may reinforce comorbidity between depression and chronic refractory migraine. Therefore, we used BDI scores .The PSQI was developed by Buysse et al. It provides a quantitative measurement of sleep quality to identify good and poor sleep. We wanted to evaluate sleep quality in our patients because chronic pain negatively affects sleep quality .These scoring concepts were used preintervention, and at the post interventional 1st and 3rd months. Afterward, whether the patients benefited from the intervention was assessed by subtracting the preintervention score from the post interventional 1st-month score, and the pre intervention score from the post interventional 3rd-month score. Demographic data of all patients, the side of the pain, and the monthly attack frequency and duration were noted.

The treatment was performed in the local operating room under sterile conditions, accompanied by ultrasonographic imaging with a linear probe (6-12-Mhz Philips DC7 color Doppler ultrasound machine), in the prone position, at the C2 level, with the head slightly flexed. No sedation is needed for this intervention.We start visualizing from the occipital protrusion,then we slide the probe inferiorly to find the first bifid spinous process of C2. After finding the C2 level, we move the probe laterally (towards the side where we will use the RF) to identify the obliquus capitis inferior muscle and semispinalis capitis muscle of the neck .The GON is found superficial to the obliquus capitis inferior muscle and deeperto the semispinalis capitis muscle at this level. After identifying the GON, a catheter needle (22-gauge 5 cm 5 mm active tip hybrid electrode) is inserted with an in-plane technique from lateral to medial. After visualizing the electrode tip placed close to the right or left GON, a sensory stimulation test is performed using an RF generator . After the patient reports dysesthesia and a tingling sensation at the occipital area with less than 0.2 V, the Pulsed RF treatment is administered at 5 Hz and 5 milliseconds pulsed width for 360 seconds at 45 V under the constraint that the temperature of the electrode tips does not exceed 42°C

ELIGIBILITY:
Inclusion Criteria:

Chronic refractory migraine patients

Exclusion Criteria:

Other primer headache disorders, İntracranial lesion, Bleeding disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this study, 25 patients who were diagnosed as having chronic refractory migraine and were refractory to conventional treatments, such as oral medications, GONB,and botulinum toxin injection were evaluated.All patients received pulsed RFtherapy to the GON from the proximal (C2) level in the pain clinic between September 2020 and September 2021.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
GON pulsed radiofrequency therapy applied from the proximal level under ultrasound guidance is effective and safe. | 3 months
  The aim of our study to evaluate the clinical responses of patients with chronic migraine who underwent pulsed Radiofrequency therapy at the C2 level under ultrasound guidance.GON pulsed radiofrequency therapy applied under the guidance of ultrasound benefited all our patients and no side effects were observed.
GON pulsed radiofrequency therapy applied from the proximal level under ultrasound guidance provides positive effects on quality of life, depression and sleep. | 3 months
  GON RF treatment provided significant improvement in the scores (BDI,MIDAS, VAS and PSQI) of all patients withmigraine in our study.

CONTACTS AND LOCATIONS:
Locations (1):
- Tepecik Training and Research Hospital, Izmir, Turkey (Türkiye)